CLINICAL TRIAL: NCT06987331
Title: The Effect of Haptonomy and Conscious Awareness Applied to Pregnant Women on Prenatal Breastfeeding Self-efficacy and Infant Feeding Attitudes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Suheyla Demirtas Alpsalaz, Principal Investigator, Inonu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Inönü university, 2024/5529
Record Dates: First submitted 2025-04-26; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy
Keywords: mindfulness; pregnancy; haptonomy; infant feeding; breastfeeding self-efficacy
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomised controlled experimental research. There are two different experimental groups in the study: Haptonomy and Mindfulness groups. The researcher has haptonomy and mindfulness certificates. The minimum sample size was calculated as 40 people for each group in total (40 haptonomy, 40 mindfulness, 40 control group) in order to reach an effect size of 0.70and 0.87 power at 5% margin of error in G-Power 3.1.9.4 programme. The data were collected by the researcher at the ASM. Haptonomy and Mindfulness practices were conducted twice a week for 4 weeks with a total of eight 30-minute interviews. Pregnant women in the experimental group were met at the first encounter and filled out the Infant Feeding Attitude Scale and Prenatal Breastfeeding Self-Efficacy Scale and Pregnant Information Form as pre-tests and post-tests were performed after the training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The effect of haptonomy and mindfulness applied to pregnant women on breastfeeding and infant nutrit (Experimental): Haptonomy and mindfulness were applied to pregnant women in two of the three groups as two experimental and one control group.
  Interventions: Other: haptonomy; Behavioral: Haptonomy application; Behavioral: Mindfulness

INTERVENTIONS:
Other: haptonomy — Haptonomy involves a combination of skills taught in 4-8 sessions of 45-60 minutes between 20 and 36 weeks of gestation. An important stage of the three-step haptonomy application is the attachment of the parents to the foetus by touching the foetus in the 20-36th weeks of pregnancy.
  Mindfullnes is a mbsr application done in 8 sessions
Behavioral: Haptonomy application — breastfeeding status
Behavioral: Mindfulness — breastfeeding status

SUMMARY:
Breast milk is an invaluable source of infant nutrition and has numerous benefits for mother and infant . Despite the benefits of breastfeeding, breastfeeding rates remain well below the level recommended by the World Health Organisation. According to the Turkish Demographic and Health Survey (TDHS) 2018 data, only 41% of infants younger than six months are breastfed and this rate decreases rapidly after the sixth month. World Health Organization (WHO), UNICEF (United Nations Children's Fund) data and studies indicate that mothers should be supported in breastfeeding and breastfeeding rates are insufficient . In order for breastfeeding rates to reach the desired level, the updated WHO guidelines on breastfeeding state that 'counselling should be provided to pregnant women and their families about the benefits and management of breastfeeding in places where antenatal care is provided' . There are many studies showing that education and training related with breastfeeding have positive effects on mothers' desire to breastfeed, breastfeeding self-efficacy, frequency of breastfeeding problems, early initiation of breastfeeding, and increased duration of breastfeeding . It has been reported that breastfeeding trainings are effective in the cognitive process and the increase in the cognitive development of women positively affects breastfeeding .

It is known that some alternative medicine methods such as music therapy, relaxation exercises and hypnosis applied during pregnancy are beneficial in breastfeeding . Haptonomy is one of the relaxation methods used in the prenatal period and is based on touching for healing. This method, which aims to develop a more positive attitude towards pregnancy and birth, is an approach in which the body and mind are considered as a whole. In general, haptonomy can be defined as a method based on body-affect-mind integrity . In the literature, it has been reported that haptonomy provides faster and easier establishment of the bond between mother, father and baby and also plays an important role in reducing birth-related complications and postpartum problems . In studies, it has been reported that haptonomy is effective in increasing the level of prenatal attachment and acceptance of pregnancy, increases the level of attachment to their babies in pregnant women and reduces the fear of birth(. It is known that haptonomy practice supports the mother's adaptation to pregnancy, psychological preparation for birth and transition to parenthood. It is also emphasised that it plays an important role in terms of psycho-physical comfort of the baby. It has been reported that haptonomy is beneficial for parents, baby and family and has a supportive effect on the practices of midwives, nurses and other health professionals . When the national and international literature is analysed, it is stated that there are not enough scientific studies despite the benefits of haptonomy .

Another method used during pregnancy is mindfulness. Mindfulness is an old Buddhist approach and its simplest definition is the art of living consciously and is defined as a type of meditation that improves the individual's ability to focus on what is happening in an accepting way . In a meta-analysis study, it was reported that mindfulness-based interventions may be useful for mindfulness levels in the perinatal period . It was reported that mindfulness interventions applied by nurses to improve maternal outcomes in pregnancy education classes had positive effects on maternal well-being . AIt is reported that the care of pregnant women is beneficial for the baby's health. . In the literature, there are many studies on the effects of mindfulness on pregnant women and newborns .

Prenatal maternal well-being has a significant effect on both mother and foetus. Therefore, it is of great importance to develop and evaluate strategies and interventions to increase well-being. Nurses' integration of mindfulness and haptonomy practices into patient care and education may positively affect women's health outcomes. In order to support the independent roles of nurses, these practices should be included in routine pregnancy and postpartum period trainings. In the literature, no study comparing haptonomy and mindfulness during pregnancy was found. However, the use of these practices in the prenatal period may contribute to the reduction of problems that may be encountered in the postpartum period and to the increase in maternal well-being. As a result, breastfeeding and infant feeding attitudes may also be positively affected and this study was planned.

ELIGIBILITY:
Inclusion Criteria:

* No verbal communication problems
* Not being diagnosed with psychological illness
* A singleton and viable pregnancy,
* No recognised pregnancy-related risk (such as pre-eclampsia, diabetes, heart disease, placenta previa, oligohydramnios),
* The fetus does not have any diagnosed health problems (such as fetal anomaly, intrauterine growth retardation)

Exclusion Criteria:

* Conceived with assisted reproductive techniques,
* Less than 20 weeks and >32 weeks of gestation
* Existing chronic disease history

Ages: 18 Months to 48 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — applied to pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
the effect of haptonomy and mindfulness applied to pregnant women on prenatal breastfeeding self-efficacy and infant feeding attitude | 8 WEEK
  prenatal breastfeeding self-effıcacy scale
  It was developed by Wells et al. (2006) to determine the breastfeeding self-efficacy perceptions of pregnant women in the prenatal period. The validity and reliability study of the scale in Turkish was conducted by Aydın and Pasinlioglu (2018) and the Cronbach's alpha coefficient of the scale was 0.85. The scale consists of a total of 20 items and four subgroups. These are; general information (items 1, 2, 3, 5, 17), skills and demands (items 6, 7, 8, 9, 10, 11, 12, 20), breastfeeding and relationship with other people (items 13, 14, 15, 16) and social pressure (items 4, 18, 19). Each item of the scale was graded on a 5-point Likert scale, where 1=Not sure at all, 2=Somewhat sure, 3=Quite sure, 4=Very sure, 5= Absolutely sure. The lowest score that can be obtained from the total scale is 20 and the highest score is 100. A high score indicates high breastfeeding self-efficacy.

SECONDARY OUTCOMES:
the effect of haptonomy and mindfulness applied to pregnant women on prenatal breastfeeding self-efficacy and infant feeding attitude | 8 week
  Iowa Infant Feeding Attitude Scale
  Infant Feeding Attitude Scale The scale developed by De La Mora and Russell was designed to evaluate women's attitudes towards breastfeeding and to determine the duration of breastfeeding as well as the choice of infant feeding method. On a five-point Likert scale, 9 items assess breastfeeding and 8 items assess formula feeding. The items evaluating formula feeding are reverse scored. The total score obtained from the scale ranges from 17 (reflects positive attitude towards bottle feeding) to 85 points (reflects positive attitude towards breastfeeding). High scores indicate a favourable breastfeeding attitude. The Turkish validity and reliability study of the scale was conducted and the cronbach alpha value was 0.71. Apart from the application of the scale in the clinic, it is recommended to be used in both antenatal and postnatal periods.

CONTACTS AND LOCATIONS:
Overall Officials: Demirtaş Alpsalaz, Principal Investigator — Bağlı Olmayan
Locations (1):
- Akdağmadeni state hospital, Yozgat, Akdağmadeni, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The effect of haptonomy and mindfulness applied to pregnant women on prenatal breastfeeding self-efficacy and infant feeding attitude
Supporting Information: Study Protocol
Time Frame: december 2025-2026
Access Criteria: users
URL: https://clinicaltrials.gov/

REFERENCES:
- See also: Related Info — https://www.ibm.com/support/pages/downloading-ibm-spss-amos-24
- Available data/document: Statistical Analysis Plan — https://www.ibm.com/support/pages/downloading-ibm-spss-amos-24 — https://www.ibm.com/support/pages/downloading-ibm-spss-amos-24